CLINICAL TRIAL: NCT06664879
Title: ALLG AMLM26 INTERCEPT (Investigating Novel Therapy to Target Early Relapse and Clonal Evolution as Pre-emptive Therapy in AML): A Multi-arm, Precision-based, Recursive, Platform Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Australasian Leukaemia and Lymphoma Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1117; NCI-2024-10306 (Other: NCI-CTRP Clinical Trial Registray)
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: AML
MeSH Terms: interventions — sabatolimab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with MBG453 + Azacitidine (Experimental): Participants will be randomized to arm
  Interventions: Drug: MBG-453 + Azacitidine

INTERVENTIONS:
Drug: MBG-453 + Azacitidine — Given intravenously (by vein)

SUMMARY:
To demonstrate the efficacy of targeted and tailored sequential therapy in patients with AML.

DETAILED DESCRIPTION:
Primary Objective:

To determine the MRD response of patients with AML to decision-rule guided therapy.

Secondary Objectives:

To determine the durability of the response of patients with AML to decision-rule guided therapy.

A key scientific objective of the study is to investigate the dynamics of MRD response and the duration of clinical benefit in the morphologic and MRD failure strata.

To investigate if duration of MRD response is longer for patients treated at MRD vs morphologic failure. Safety: To characterize the safety and tolerability of targeted therapies (as single agents and in combination with other agents).

To investigate the efficacy of distinct treatment sequences in AML patients who fail one or more lines of therapy on study.

To determine the overall efficacy of the platform as an evolving system for managing patients with AML. Quality of Life.

To investigate patterns and mechanisms of resistance.

To determine the response of patients with AML with morphologic relapse in each treatment arm.

To determine the response of patients with AML with a secondary MRD marker in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Meets inclusion criteria outlined in the AMLM26 INTERCEPT Master Protocol including:

   1. Master Protocol Inclusion Criteria listed in Master Protocol Appendix 3.0.
   2. the mutation/mutations specified for this treatment arm in Master Protocol Appendix 2.0 Compendium of Actionable Domains and Allocation Rules
2. Meets MRD eligibility for INTERCEPT therapy based on a screening sample taken no more than 42 days prior to cycle 1 of day 1 of treatment on this treatment arm. Refer to Master Protocol Appendix 5 for the definitions of MRD progression/failure. Eligibility will be confirmed by the MRD review committee.
3. ECOG 0-2
4. Patients entering this arm post-allogeneic stem cell transplantation will need to have an absolute lymphocyte count of .0.2 x 109/L and no evidence of active acute graft-versushost disease (GVHD)
5. Subject must have adequate renal function as demonstrated by a creatinine clearance .

30 mL/min; calculated by the Cockcroft Gault formula or measured by 24-hours urine collection 6. Subject must have adequate liver function as demonstrated by:

1. aspartate aminotransferase (AST) . 3.0 ~ ULN
2. alanine aminotransferase (ALT) . 3.0 ~ ULN
3. bilirubin . 1.5 ~ ULN (unless bilirubin rise is due to Gilbert fs syndrome or of nonhepatic origin) 7. Agrees to follow the recommended contraception procedures for this treatment domain

Exclusion Criteria:

Presence of any general exclusion criteria outlined in the AMLM26 INTERCEPT Master Protocol 2. Prior allogeneic stem cell transplantation within 3 months of post-conditioning or on

* 10mg/day prednisolone for graft vs host disease 3. Subject is HIV positive 4. Patients with .5% myeloblasts in bone marrow on morphologic assessment 5. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  1. Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
  2. Acute/Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) or resolved HBV infection may participate. 6. Systemic chronic corticosteroid therapy (≥10 mg/day prednisone or equivalent) or any immunosuppressive therapy within 7 days of first dose of study treatment. Topical, inhaled, nasal and ophthalmic steroids are allowed. 7. For initial enrolment to INTERCEPT therapy, patients who have received previous TIM3 inhibitor treatment are excluded. This exclusion criteria does not apply to patients crossing-over from MBG453 arm to the combination MBG453 + azacitidine arm, unless MBG453 was ceased due to MBG453-related toxicity. 8. Patients with active, known or suspected autoimmune disease. Patients with vitiligo, type I diabetes, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur should not be excluded 9. History of or current drug-induced interstitial lung disease or pneumonitis grade .2 10. Subject has been diagnosed with another malignancy, unless disease-free for at least 2 years and not needing active treatment. Patients with fully excised BCC/SCC/CIN or other minor malignancy are not excluded 11. Subject has clinically significant abnormality of coagulation profile, such as disseminated intravascular coagulation 12. Use of any live vaccines against infectious diseases (i.e. Influenza, varicella, pneumococcus) within 4 weeks of initiation of study treatment 13. Impaired cardiac function or clinically significant cardiac disease, including any of the following:
* Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (NYHA Grade . 2) with an LVEF of <40%, uncontrolled hypertension or clinically significant arrhythmia
* Acute myocardial infarction or unstable angina pectoris . 3 months prior to study entry 14. Known hypersensitivity to azacitidine or mannitol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org